CLINICAL TRIAL: NCT05635669
Title: Optimized Acupuncture Treatment for Female Stress Urinary Incontinence: a Study Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Optimized Acupuncture Treatment for Female Stress Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yin Ping (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Sponsor-Investigator, Yin Ping, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22Y21920100
Record Dates: First submitted 2022-11-12; First posted 2022-12-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sacral acupoints group (Sacral group) (Experimental): Participants will receive sacral acupoints combination treatment at bilaterally Huiyang(BL35) and Zhongliao(BL33) with prone position during the whole treatment course.
  Interventions: Device: Sacral acupoints acupuncture
- Abdominal acupoints group (Abdominal group) (Experimental): Participants will receive abdominal acupoints combination treatment at unilateral Zhongji(RN3), Guanyuan(RN4) and bilaterally Dahe(KI12) with dorsal position during the whole treatment course.
  Interventions: Device: Abdominal acupoints acupuncture
- Alternating acupoints group (Alternating group) (Experimental): Participants will receive treatment of sacral acupoints combination and abdominal acupoints combination alternately. (For example, A for the first time, B for the second time, A for the third time, and so on. )
  Interventions: Device: Alternating acupoints acupuncture

INTERVENTIONS:
Device: Sacral acupoints acupuncture — Before treatment, the participants will be asked to go to the toilet. All treatments will be performed after skin disinfection. As acupuncture needles are inserted, all points will be lifted, twisted, and stabbed to activate the sensation of de qi. The electroacupuncture stimulation lasted for 30 minutes with a continuous wave of 50 Hz and a current intensity of 1 to 5 mA (preferably with the skin around the acupoints shivering mildly without pain). Participants will receive three treatments per week (every other day), each lasting 30 minutes, for a total of 18 sessions over the course of 6 weeks. The follow-up sessions are on week 18, 30, 42 and 54. In this group, paired electrodes from the electroacupuncture apparatus were attached transversely to the needle handles at bilateral Huiyang(BL35) and Zhongliao(BL33) .
  Arms: Sacral acupoints group (Sacral group)
Device: Abdominal acupoints acupuncture — Before treatment, the participants will be asked to go to the toilet. All treatments will be performed after skin disinfection. As acupuncture needles are inserted, all points will be lifted, twisted, and stabbed to activate the sensation of de qi. The electroacupuncture stimulation lasted for 30 minutes with a continuous wave of 50 Hz and a current intensity of 1 to 5 mA (preferably with the skin around the acupoints shivering mildly without pain). Participants will receive three treatments per week (every other day), each lasting 30 minutes, for a total of 18 sessions over the course of 6 weeks. The follow-up sessions are on week 18, 30, 42 and 54. In this group, paired electrodes from the electroacupuncture apparatus were attached to the needle handles respectively at Zhongji(RN3) and one side of Dahe(KI12), as well as Guanyuan(RN4) and another side of Dahe(KI12).
  Arms: Abdominal acupoints group (Abdominal group)
Device: Alternating acupoints acupuncture — Before treatment, the participants will be asked to go to the toilet. All treatments will be performed after skin disinfection. As acupuncture needles are inserted, all points will be lifted, twisted, and stabbed to activate the sensation of de qi. The electroacupuncture stimulation lasted for 30 minutes with a continuous wave of 50 Hz and a current intensity of 1 to 5 mA (preferably with the skin around the acupoints shivering mildly without pain). Participants will receive three treatments per week (every other day), each lasting 30 minutes, for a total of 18 sessions over the course of 6 weeks. The follow-up sessions are on week 18, 30, 42 and 54. The application of electroacupuncture is the same as Sacral group and Abdominal group.
  Arms: Alternating acupoints group (Alternating group)

SUMMARY:
This multicenter randomized controlled trial is designed to explore a relatively suitable application of acupoint combinations and to provide certain clinical evidence for the optimization of acupuncture treatment of female SUI.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) mainly refers to the involuntary leakage of urine when abdominal pressure increases, such as sneezing, coughing, laughing or exercise. According to epidemiological studies, the global median prevalence of female urinary incontinence is 27.6% (4.8%-58.4%), of which SUI accounts for more than 50%. Previous study have demonstrated that acupuncture intervention can reduce the urine leakage in pad test, decrease the ICIQ-SF score, so as to help the patients alleviate the symptoms and improve their quality of life. This multicenter randomized controlled trial set 3 groups. Patients will receive 3 different applications of acupoint combinations so that the optimization of acupuncture treatment of female SUI will be find.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate SUI mentioned in the diagnostic criteria above;
* Aged 40～75 years;
* Sign the informed consent.

Exclusion Criteria:

* Other types of urinary incontinence (urgent, overflow or mixed).
* History of urinary incontinence surgery or pelvic floor surgery;
* Pelvic organ prolapse ≥ stage II;
* Symptomatic urinary tract infection;
* Residual urine volume > 30 mL;
* Maximum urinary flow rate < 20ml/s.
* Limitation of movement (walk and/or run and/or climb stairs);
* Patients who have been using drugs that may affect bladder function or receiving SUI specialized treatment;
* Severe cardiovascular, cerebral, liver, kidney and hematopoietic system disease, mental disorders, diabetes, multiple system atrophy, cauda equina neuropathy and spinal cord disease;
* Pregnancy or lactation period.
* With cardiac pacemaker, acupuncture phobia or metal allergies;

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The change of urine leakage measured by the 1-hour pad test | Week 6
  Quantity of fluid loss will be measured by 1-hour pad test, compared with the baseline (week 0).

SECONDARY OUTCOMES:
The change of mean episodes of urinary incontinence in 72 hours | Week 4, 6, 18, 30, 42 and 54
  The mean episodes of urinary incontinence in 72 hours based on '72 hours bladder diary', comparing the value at week 4, 6, 18, 30, 42 and 54 with the baseline(week 0).
The change of International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Week 4, 6, 18, 30, 42 and 54
  ICIQ-SF is a brief instrument used to assess the frequency of incontinence, the volume of incontinence, as well as the impact of life quality). The value will be recorded at week 4, 6, 18, 30, 42 and 54, compared to that at baseline(week 0).
Severity of SUI according to '72 hours bladder diary' | Week 4, 6, 18, 30, 42 and 54
  The severity of SUI will be rated according to the amount of UI in usual conditions without extreme activities like severe cough, strenuous exercise or carrying heavy loads in the past 72 hours. Definition: mild(several drops of leakage);moderate(leak that soaked through underwear); severe(leak that soaked through outerwear). In case that participants worn urinal pads, the severity of SUI will be graded as follows. Mild(several drops of leakage); moderate(soaked urine pads in patches by several leakages); severe(soaked urine pads in patches by one leakage). The most severe degree of urine leakage in patient's 72 hours bladder diaries over the assessment period will be selected as the severity of SUI for analyses.
Participant Self-evaluation of Therapeutic Effects | Week 4, 6, 18, 30, 42 and 54
  No help=0; Small help=1; Medium help=2; Great help=3
The number of patients who used other treatment for SUI | Week 18, 30, 42 and 54
  Compare the number of patients who used other specialty therapy for SUI during the study between 3 groups.
Bladder neck mobility by pelvic floor ultrasonography | Week 6
  Bladder neck mobility will be observed both at rest and during a Valsalva maneuver by pelvic floor ultrasonography. The result can be measured from the ultrasonic image.
Urethral rotation angle by pelvic floor ultrasonography | Week 6
  Urethral rotation angle will be observed both at rest and during a Valsalva maneuver by pelvic floor ultrasonography. The result can be measured from the ultrasonic image.
Retrovesical angle by pelvic floor ultrasonography | Week 6
  Retrovesical angle will be observed both at rest and during a Valsalva maneuver by pelvic floor ultrasonography. The result can be measured from the ultrasonic image.
Lowest point of bladder by pelvic floor ultrasonography | Week 6
  Lowest point of bladder at rest and during a Valsalva maneuver by pelvic floor ultrasonography. The result can be observed from the ultrasonic image.
Urethral funnel formation by pelvic floor ultrasonography | Week 6
  Urethral funnel formation at rest and during a Valsalva maneuver by pelvic floor ultrasonography. The result can be observed from the ultrasonic image.
The type of bladder bulging by pelvic floor ultrasonography | Week 6
  The type of bladder bulging at rest and during a Valsalva maneuver by pelvic floor ultrasonography. The result can be observed from the ultrasonic image.
Subgroup analysis: correlation between 1-hour pad test and severity of SUI | Week 6
  Analyze the correlation between 1-hour pad test and severity of SUI.
Subgroup analysis: correlation between episodes of urinary incontinence in 72 hours and severity of SUI | Week18, 30, 42 and 54
  Analyze the correlation between episodes of urinary incontinence in 72 hours and severity of SUI.
Number of urine pads used weekly | Week 4, 6, 18, 30, 42 and 54
  The weekly consumption of urine pads was assessed in participants.
Incidence of adverse events | Week 1-6
  Observe the incidence of adverse events during the treatment.
Evaluation of discomfort during treatment | Within 5 minutes after the first and ninth acupuncture treatment
  Visual analog scale (VAS) will be used to evaluate the degree of discomfort during treatment. The scale ranging from 0 to 10cm, with 0cm indicating no discomfort and 10cm indicating severe discomfort. Evaluation time: The average value of the first and ninth acupuncture treatments was taken within 5 minutes after the end of the two treatments. If the VAS value is missing in one of the cases, another is taken as the result.
Patient acceptability evaluation | Within 5 minutes after the first and ninth acupuncture treatment
  0=very difficult to accept, 1=slightly difficult to accept, 2=acceptable, 3=easy to accept, 4=very easy to accept. Evaluation time: The average value of the first and ninth acupuncture treatments was taken within 5 minutes after the end of the two treatments. If the VAS value is missing in one of the cases, another is taken as the result.

CONTACTS AND LOCATIONS:
Overall Officials: YUELAI CHEN, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang N, Ge X, Ye J, Liu Q, Wu Y, Yan H, Han X. Efficacy of acupuncture for urinary incontinence in middle-aged and elderly women: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2021 Feb;257:138-143. doi: 10.1016/j.ejogrb.2020.11.001. Epub 2020 Nov 4. PMID 33419589
- [Background] Liu Z, Liu Y, Xu H, He L, Chen Y, Fu L, Li N, Lu Y, Su T, Sun J, Wang J, Yue Z, Zhang W, Zhao J, Zhou Z, Wu J, Zhou K, Ai Y, Zhou J, Pang R, Wang Y, Qin Z, Yan S, Li H, Luo L, Liu B. Effect of Electroacupuncture on Urinary Leakage Among Women With Stress Urinary Incontinence: A Randomized Clinical Trial. JAMA. 2017 Jun 27;317(24):2493-2501. doi: 10.1001/jama.2017.7220. PMID 28655016
- [Background] Nambiar AK, Arlandis S, Bo K, Cobussen-Boekhorst H, Costantini E, de Heide M, Farag F, Groen J, Karavitakis M, Lapitan MC, Manso M, Arteaga SM, Riogh ANA, O'Connor E, Omar MI, Peyronnet B, Phe V, Sakalis VI, Sihra N, Tzelves L, van Poelgeest-Pomfret ML, van den Bos TWL, van der Vaart H, Harding CK. European Association of Urology Guidelines on the Diagnosis and Management of Female Non-neurogenic Lower Urinary Tract Symptoms. Part 1: Diagnostics, Overactive Bladder, Stress Urinary Incontinence, and Mixed Urinary Incontinence. Eur Urol. 2022 Jul;82(1):49-59. doi: 10.1016/j.eururo.2022.01.045. Epub 2022 Feb 23. PMID 35216856
- [Background] Guan LX, Song XL, Wang X, Zhang X, Liu LM, Chen BL, Chen YL. Immediate effects of Zhongji point acupuncture on pelvic floor structure in female patients with stress urinary incontinence: a randomized, single-blind, and sham-controlled clinical trial protocol. Ann Palliat Med. 2021 Jul;10(7):8292-8299. doi: 10.21037/apm-21-662. Epub 2021 Jul 2. PMID 34263647
- [Derived] Liu L, Chen B, Si X, Hou W, Fan Q, Li X, Li J, Ming S, Yin P, Chen Y. Optimized electroacupuncture treatment for female stress urinary incontinence: study protocol for a multi-center randomized controlled trial. Front Psychiatry. 2023 Aug 17;14:1228131. doi: 10.3389/fpsyt.2023.1228131. eCollection 2023. PMID 37663593